CLINICAL TRIAL: NCT05037539
Title: Efficacy of Injectable Fentanyl in Sublingual Route Versus Oral Morphine Syrup for Breakthrough Pain in Gynecologic Cancer Patients With Chronic Cancer Pain : A Randomized Double Blind Controlled Trial
Brief Title: Efficacy of Injectable Fentanyl in Sublingual Route Versus Oral Morphine Syrup for Breakthrough Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 090/2564
Record Dates: First submitted 2021-05-24; First posted 2021-09-08 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2021-08

CONDITIONS: Pain, Breakthrough
Keywords: breakthrough pain; Injectable Fentanyl in Sublingual Route; gynecologic cancer
MeSH Terms: conditions — Breakthrough Pain | interventions — Fentanyl; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injectable Fentanyl in Sublingual Route (Experimental): Injectable Fentanyl in Sublingual Route that given after the first time Breakthrough Pain is occurred 50 mcg in sublingual route
  Interventions: Drug: Fentanyl Citrate 50Mcg/Ml Inj_#1
- Oral Morphine Syrup (Active Comparator): Oral Morphine Syrup 2.5 ml ( 5 mg) in oral router that first time given after Breakthrough Pain is occurred
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl Citrate 50Mcg/Ml Inj_#1 — Injectable Fentanyl in Sublingual Route 50 mcg
  Other Names: Fentanyl
  Arms: Injectable Fentanyl in Sublingual Route
Drug: Morphine — Oral Morphine Syrup 2.5 ml ( 5 mg)
  Other Names: morphine syrup
  Arms: Oral Morphine Syrup

SUMMARY:
Randomized control trial that to comparison the efficacy of injectable fentanyl in sublingual route versus oral morphine syrup for breakthrough pain in gynecologic cancer patients with chronic cancer pain Primary outcome : to measure pain score after drug is given

DETAILED DESCRIPTION:
objective; To comparison the efficacy of injectable fentanyl in sublingual route versus oral morphine syrup for breakthrough pain in gynecologic cancer patients with chronic cancer pain Population : gynecologic cancer patients with chronic cancer pain that use opioid drug for basal pain and had experienced of breakthrough pain cancer in Rajavithi hospital sample size : 20 person/group Method ; Randomized control trial , Prospective Intervention : group A : injectable fentanyl in sublingual , group B : oral morphine syrup Primary outcome : to measure pain score after drug is given at 5, 15, 30, 45, 60 and 120 min secondary outcome : to record side effect of drug is given at 5, 15, 30, 45, 60 and 120 min Statistical method

* Categorical data = Chi-square test or Fishers' exact test
* Continuous data : comparison with Student t-test in normal deviation data and Man-Whitney U- test in abnormal deviation data • Analytical data with Pearson's correlation, Linear regression or Binary Logistic regression, Repeated Measures ANOVA with OR (95%CI) and p-value <0.05

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer patients with chronic cancer pain that use opioid drug for basal pain

Exclusion Criteria:

* allergy in fentanyl or morphine
* abnormal cognitive function patient

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pain score | after drug is given at 5 minutes
  measure with numeric score from 0-10 point (maximum pain= 10 point)

SECONDARY OUTCOMES:
Neausea and vomiting | after drug is given at 5 minutes
  measure by asking symptom from patient
Ithching | after drug is given at 5 minutes
  measure by asking symptom from patient
Respiratory distress | after drug is given at 5 minutes
  measure by respiratory rate parametor

CONTACTS AND LOCATIONS:
Overall Officials: Thanvarat Tilagul, Study Director — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lennernas B, Hedner T, Holmberg M, Bredenberg S, Nystrom C, Lennernas H. Pharmacokinetics and tolerability of different doses of fentanyl following sublingual administration of a rapidly dissolving tablet to cancer patients: a new approach to treatment of incident pain. Br J Clin Pharmacol. 2005 Feb;59(2):249-53. doi: 10.1111/j.1365-2125.2004.02264.x. PMID 15676050
- [Result] Portenoy RK, Payne D, Jacobsen P. Breakthrough pain: characteristics and impact in patients with cancer pain. Pain. 1999 May;81(1-2):129-34. doi: 10.1016/s0304-3959(99)00006-8. PMID 10353500
- [Result] Zeppetella G. Opioids for cancer breakthrough pain: a pilot study reporting patient assessment of time to meaningful pain relief. J Pain Symptom Manage. 2008 May;35(5):563-7. doi: 10.1016/j.jpainsymman.2007.06.012. Epub 2008 Feb 6. PMID 18258412
- [Result] Mercadante S. The use of rapid onset opioids for breakthrough cancer pain: the challenge of its dosing. Crit Rev Oncol Hematol. 2011 Dec;80(3):460-5. doi: 10.1016/j.critrevonc.2010.12.002. Epub 2011 Jan 6. PMID 21215653
- [Result] Jandhyala R, Fullarton JR, Bennett MI. Efficacy of rapid-onset oral fentanyl formulations vs. oral morphine for cancer-related breakthrough pain: a meta-analysis of comparative trials. J Pain Symptom Manage. 2013 Oct;46(4):573-80. doi: 10.1016/j.jpainsymman.2012.09.009. Epub 2013 Feb 4. PMID 23380337
- [Result] Velazquez Rivera I, Munoz Garrido JC, Garcia Velasco P, Espana Ximenez de Enciso I, Velazquez Clavarana L. Efficacy of sublingual fentanyl vs. oral morphine for cancer-related breakthrough pain. Adv Ther. 2014 Jan;31(1):107-17. doi: 10.1007/s12325-013-0086-4. Epub 2014 Jan 3. PMID 24385406
- [Result] Bushnaq M, Al-Shoubaki M, Milhem M. The feasibility of using intravenous fentanyl as sublingual drops in the treatment of incidental pain in patients with cancer. J Palliat Med. 2009 Jun;12(6):511-4. doi: 10.1089/jpm.2009.9618. No abstract available. PMID 19508134
- [Derived] Thantiprechapong T, Tilagul T, Vasikasin V. Efficacy of reconstituted intravenous fentanyl to sublingual solution versus oral morphine syrup for breakthrough pain among patients with chronic gynecologic cancer pain: A randomized, double-blind, placebo-controlled trial. J Obstet Gynaecol Res. 2023 Jul;49(7):1815-1820. doi: 10.1111/jog.15674. Epub 2023 May 11. PMID 37170709